CLINICAL TRIAL: NCT02436629
Title: The Effect of Nitrate Supplementation on Sport Performance: High Intensity Intermittent Performance in Recreational Athletes
Brief Title: Nitrate for High Intensity Intermittent Exercise
Acronym: NITR-ITE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: METC 153006
Record Dates: First submitted 2015-05-04; First posted 2015-05-07 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-03

CONDITIONS: High Intensity Intermittent Sports Performance
Keywords: Red beetroot juice; High intensity intermittent exercise; Nitrite; Soccer

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nitrate-rich concentrated beetroot juice (Active Comparator): Dietary supplement: 800 mg of nitrate in 140 mL of concentrated beetroot juice (Beet-IT)
  Interventions: Dietary Supplement: Nitrate-rich concentrated beetroot juice
- Nitrate-depleted conc. beetroot juice (Placebo Comparator): Placebo: 140 mL of nitrate-depleted concentrated red beetroot juice
  Interventions: Dietary Supplement: Nitrate-depleted concentrated red beetroot juice

INTERVENTIONS:
Dietary Supplement: Nitrate-rich concentrated beetroot juice — James White, Beet It Sport Shot, 70ml (Standard)
  Arms: Nitrate-rich concentrated beetroot juice
Dietary Supplement: Nitrate-depleted concentrated red beetroot juice — Beet It Sport Shot, 70ml (Placebo)
  Arms: Nitrate-depleted conc. beetroot juice

SUMMARY:
The objective of the current study is to assess the effect of 6-day dietary nitrate ingestion on high intensity intermittent sports performance in recreational soccer players.

DETAILED DESCRIPTION:
Oral ingestion of nitrate (NO3-) in the form of both nitrate salts and concentrated red beetroot juice has been shown to significantly lower blood pressure at rest and to improve exercise performance during cycle time trials. Furthermore, a positive exercise performance effect of nitrate ingestion has been observed in recreational athletes during intermittent exercise. However, this was achieved after acute supplementation with a substantial dose of dietary nitrate. Whether similar ergogenic effects of nitrate supplementation can be achieved with a more conventional 6-day nitrate supplementation protocol with a lower daily dose remains to be established. Based on the gaps in current literature, our main goal will be to gain further insight into the effects of a 6-day nitrate supplementation protocol on high intensity intermittent exercise performance in recreational athletes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy P
* Players of the first two senior selection teams of a regional soccer club competing at the 3rd KNVB level or higher
* Training ≥2 days a week
* 18-40 years
* Male

Exclusion Criteria:

* Use of medication
* Injury prohibiting them from performing the exercise protocol effectively
* Smoking
* Currently supplementing diet with nitrate
* Lactose intolerance

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-05; Primary Completion 2016-04 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Total distance covered during the Yo-Yo Intermittent Recovery 1 test (Yo-Yo IR1 test) | Performance 3 hours post red beetroot juice ingestion

SECONDARY OUTCOMES:
Plasma concentration of nitrite and nitrate | Concetrations 3 hours post red beetroot juice ingestion
Salivary concentration of nitrite and nitrate | Concetrations 3 hours post red beetroot juice ingestion

OTHER OUTCOMES:
Baseline characteristics | 30 min during visit 1 (Screening)
  Height, body weight, age, BMI

CONTACTS AND LOCATIONS:
Overall Officials: Lex B Verdijk, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University Medical Centre+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wylie LJ, Mohr M, Krustrup P, Jackman SR, Ermiotadis G, Kelly J, Black MI, Bailey SJ, Vanhatalo A, Jones AM. Dietary nitrate supplementation improves team sport-specific intense intermittent exercise performance. Eur J Appl Physiol. 2013 Jul;113(7):1673-84. doi: 10.1007/s00421-013-2589-8. Epub 2013 Feb 1. PMID 23370859
- [Background] Bond H, Morton L, Braakhuis AJ. Dietary nitrate supplementation improves rowing performance in well-trained rowers. Int J Sport Nutr Exerc Metab. 2012 Aug;22(4):251-6. doi: 10.1123/ijsnem.22.4.251. Epub 2012 Jun 15. PMID 22710356
- [Background] Cermak NM, Gibala MJ, van Loon LJ. Nitrate supplementation's improvement of 10-km time-trial performance in trained cyclists. Int J Sport Nutr Exerc Metab. 2012 Feb;22(1):64-71. doi: 10.1123/ijsnem.22.1.64. PMID 22248502
- [Background] Bangsbo J, Iaia FM, Krustrup P. The Yo-Yo intermittent recovery test : a useful tool for evaluation of physical performance in intermittent sports. Sports Med. 2008;38(1):37-51. doi: 10.2165/00007256-200838010-00004. PMID 18081366